CLINICAL TRIAL: NCT04544410
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of SPR001 (Tildacerfont) in Reducing Supraphysiologic Glucocorticoid Use in Adult Subjects With Classic Congenital Adrenal Hyperplasia
Brief Title: A Ph2b to Evaluate Tildacerfont in the Reduction of Glucocorticoid Steroid Doses in Adult CAH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study did not meet its primary endpoint.
Sponsor: Spruce Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPR001-204; CAHmelia 204 (Other: Spruce Biosciences)
Record Dates: First submitted 2020-08-30; First posted 2020-09-10 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: CAH; Adrenal Disorder; Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Adrenal Gland Diseases

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 manner to either Tildacerfont or Placebo for 24 weeks followed by 52 weeks open label Tildacerfont
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind for first 24 weeks, then open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tildacerfont Group (Experimental): Tildacerfont administered daily via oral tablet for 24 weeks at dose level 1; followed by open label tildacerfont for 52 weeks
  Interventions: Drug: Tildacerfont/Placebo
- Placebo (Placebo Comparator): Placebo administered daily via oral tablet for 24 weeks; followed by open label tildacerfont for 52 weeks
  Interventions: Drug: Tildacerfont/Placebo

INTERVENTIONS:
Drug: Tildacerfont/Placebo — Tablet, administered daily
  Other Names: SPR001

SUMMARY:
An investigation of the ability of Tildacerfont to reduce supraphysiologic glucocorticoid dosing in classic Congenital adrenal hyperplasia (CAH) subjects up to 76 weeks of treatment. Optional open label extension up to 240 weeks.

DETAILED DESCRIPTION:
This is a study that evaluated the ability of tildacerfont to reduce the glucocorticoid steroid dose used by adult subjects with CAH. The first 24-weeks were a double-blind, placebo controlled, comparison of tildacerfont vs placebo. The following 52-weeks allowed all subjects to move to open label tildacerfont to continue to reduce steroid dose where appropriate, and observe long term safety. Subjects were offered a long term open label extension up to 240 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥18 years old at screening
2. Has a known childhood diagnosis of classic CAH due to 21-hydroxylase deficiency based on genetic mutation in CYP21A2 and/or documented (at any time) elevated 17-hydroxyprogesterone (17-OHP) and currently treated with hydrocortisone (HC), HC acetate, prednisone, prednisolone, methylprednisolone, dexamethasone (or a combination of the aforementioned glucocorticoid [GCs])
3. Has lower limit of detection ≤ androstenedione (A4) ≤ 2.5x upper limit of normal (ULN) at screening measured before a morning GC dose
4. Has been on a stable, supraphysiologic dose of GC replacement (defined as ≥30 mg/day and ≤60 mg/day in HCe) for ≥1 month before screening
5. For subjects with the salt-wasting form of CAH, subject has been on a stable dose of mineralocorticoid replacement for ≥1 month before screening
6. Agrees to follow contraception guidelines. Male subjects must also agree to refrain from donating sperm throughout the Treatment Period and for 90 days after the last dose of study drug
7. Is able to understand all study procedures and risks involved and provides written informed consent indicating willingness to comply with all aspects of the protocol

Exclusion Criteria:

1. Has a known or suspected diagnosis of any other known form of classic CAH (not due to 21-hydroxylase deficiency)
2. Has a history that includes bilateral adrenalectomy or hypopituitarism
3. Has a history of allergy or hypersensitivity to tildacerfont, any of its excipients, or any other CRF1 receptor antagonist
4. Shows clinical signs or symptoms of adrenal insufficiency
5. Has had a clinically significant unstable medical condition, medically significant illness, or chronic disease occurring within 30 days of screening, including but not limited to:

   1. An ongoing malignancy or <3 years of remission history from any malignancy, other than successfully treated localized skin cancer
   2. eGFR of <45 mL/min/1.73 m2
   3. Current or history of liver disease (with the exception of Gilbert's syndrome)
   4. History of alcohol or substance abuse within the last year, or any significant history of alcohol or substance abuse that would likely prevent the subject from reliably participating in the study, based on the opinion of the Investigator
   5. Active hepatitis B, hepatitis C, or HIV at screening
   6. Subjects who plan to undergo bariatric surgery during the study are excluded
   7. Any other condition that would impact subject safety or confound interpretation of study results
6. Psychiatric conditions, including but not limited to bipolar disorder, schizophrenia, or schizoaffective disorders that are not effectively controlled on medication and may have an adverse impact on study compliance. Symptoms including hallucinations, delusions, and psychosis are exclusionary. Additionally:

   Increased risk of suicide based on the Investigator's judgment or the results of the C-SSRS conducted at screening and baseline (eg, C-SSRS Type 3, 4, or 5 ideation within the past 6 months or any suicidal behavior within the past 12 months) b. Hospital Anxiety and Depression Scale (HADS) score >12 for either depression or anxiety at screening or baseline
7. Has clinically significant abnormal ECG or clinical laboratory results. Abnormal results that must be reviewed and discussed with the Medical Monitor to determine eligibility for this study include but are not limited to:

   1. Any clinically meaningful abnormal ECG results, including QTcF >450 ms for male participants or >470 ms for female participants
   2. ALT >2x ULN
   3. Total bilirubin >1.5x ULN
   4. Total bile acids >5x ULN
8. Routinely works overnight shifts
9. Subjects with travel plans/work schedules that result in significant and frequent changes in time zones (>2 hours) will require Medical Monitor approval for enrollment
10. Females who are pregnant or nursing
11. Use of any other investigational drug from 30 days or 5 half-lives (whichever is longer) before screening to the end of the study
12. Use of the following drugs from 30 days or 5 half-lives (whichever is longer) before the start of the Treatment Period to the end of the study:

    1. Rosiglitazone, aromatase inhibitors, testosterone, growth hormones, or any other medication or supplement that could impact subject safety or confound interpretation of study results
    2. The drugs which are:

    i. Moderate to strong inhibitors and/or inducers of CYP3A4 ii. Sensitive substrates or narrow-therapeutic-range substrates of CYP3A4 (except hormonal contraception containing ≤35 μg ethinyl estradiol) iii. Sensitive substrates or narrow-therapeutic-range substrates of BCRP (except those that can be administered QD in the morning, separated by approximately 10 hours from evening administration of study drug)
13. Donation or receipt of blood from 90 days before Screening to the end of the study; donation or receipt of platelets, white blood cells, or plasma from 30 days before Screening to the end of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Newfield, M.D, Principal Investigator — Rady Children's Hospital-San Diego and Professor of clinical pediatrics at UC San Diego School of Medicine.
Locations (41):
- United States (16):
  - Spruce Study Site, Birmingham, Alabama
  - Spruce Study Site, Los Angeles, California
  - Spruce Study Site, San Diego, California
  - Spruce Study Site, Indianapolis, Indiana
  - Spruce Study Site, Baltimore, Maryland
  - Spruce Biosciences Clinical Site, Ann Arbor, Michigan
  - Spruce Study Site, Minneapolis, Minnesota
  - Spruce Study Site, New Brunswick, New Jersey
  - Spruce Study Site, Canton, Ohio
  - Spruce Study Site, Cincinnati, Ohio
  - Spruce Study Site, Cleveland, Ohio
  - Spruce Study Site, Columbus, Ohio
  - Spruce Study Site, Philadelphia, Pennsylvania
  - Spruce Study Site, Providence, Rhode Island
  - Spruce Study Site, Columbia, South Carolina
  - Spruce Study Site, Fort Worth, Texas
- Australia (4):
  - Spruce Study Site, Blacktown
  - Spruce Study Site, Brisbane
  - Spruce Study Site, Elizabeth Vale
  - Spruce Study Site, Parkville
- Brazil (2):
  - Spruce Study Site, Curitiba
  - Spruce Study Site, São Paulo
- Canada (2):
  - Spruce Study Site, Ottawa, Ontario
  - Spruce Study Site, Sherbrooke, Quebec
- Estonia (2):
  - Spruce Study Site, Tallinn
  - Spruce Study Site, Tartu
- Spruce Study Site, Munich, Germany
- Spruce Study Site, Roma, Italy
- Spruce Study Site, Riga, Latvia
- Spruce Study Site, Kaunas, Lithuania
- Poland (2):
  - Spruce Study Site, Krakow
  - Spruce Study Site, Warsaw
- Spruce Study Site, Bucharest, Romania
- Spruce Study Site, Seoul, South Korea
- Spain (4):
  - Spruce Study Site, Barcelona
  - Spruce Study Site, Madrid
  - Spruce Study Site, Seville
  - Spruce Study Site, Tarragona
- Spruce Study Site, Stockholm, Sweden
- Spruce Study Site, Istanbul, Turkey (Türkiye)
- Spruce Study Site, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study randomized approximately 100 participants with classic congenital adrenal hyperplasia (CAH) currently receiving glucocorticoid (GC) at a supraphysiologic dose
Pre-assignment Details: An optional Screening visit to capture information within 45 days of Day 1 in this study may have been used to determine eligibility and fulfill screening requirements for this study.
  A 6- or 12 week GC Conversion Period (Week -12 to either Week -6 or Week -2 [±3 days]) for participants on dexamethasone at the initial Screening Visit who agreed to convert to a non-dexamethasone regimen as determined by their physician.
Groups:
- Tildacerfont Group: Tildacerfont 200 mg administered daily via oral tablet for 24 weeks; followed by open label tildacerfont 200 mg for 52 weeks
- Placebo: Placebo administered daily via oral tablet for 24 weeks; followed by open label tildacerfont 200 mg for 52 weeks
Period: Double-blind Treatment Period
Arm/Group | Tildacerfont Group | Placebo
Started | 48 | 52
Completed | 44 | 50
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Open-Label Treatment Period
Arm/Group | Tildacerfont Group | Placebo
Started | 42 | 50
Completed | 20 | 24
Not Completed | 22 | 26
Not completed — Study Terminated | 15 | 19
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tildacerfont Group | Placebo | Total
Number analyzed (Participants) | 48 | 52 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (11.52) | 32.0 (12.08) | 32.5 (11.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 53
  Male | 23 | 24 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 41 | 44 | 85
  Unknown | 0 | 2 | 2
  Asian | 6 | 8 | 14
  Black or African American | 3 | 0 | 3
  White | 38 | 43 | 81
  Other | 1 | 1 | 2
Females with Child-Bearing Potential [Count of Participants; unit: Participants] | 22 | 26 | 48
Time Since Congenital adrenal hyperplasia (CAH) Diagnosis [Mean (Standard Deviation); unit: years] | 31.2 (11.58) | 28.0 (12.99) | 29.5 (12.37)
Type of CAH Diagnosis [Count of Participants; unit: Participants]
  Salt-wasting | 36 | 35 | 71
  Simple Virilizing | 12 | 17 | 29
17-hydroxyprogesterone (17-OHP) [Mean (Standard Deviation); unit: ng/dL] | 5642.5 (7481.57) | 5656.6 (6995.03) | 5649.8 (7195.84)
Androstenedione (A4) [Mean (Standard Deviation); unit: ng/dL] | 227.2 (247.10) | 222.2 (203.28) | 224.6 (224.24)
Adrenocorticotropic hormone, corticotropin (ACTH) [Mean (Standard Deviation); unit: pg/mL] | 176.79 (316.658) | 159.77 (190.594) | 167.94 (257.663)
Testosterone [Mean (Standard Deviation); unit: ng/dL] — Population: 1 participant did not have the testosterone assessment completed at baseline and this was noted as a protocol deviation
  ng/dL
    number analyzed (Participants) | 47 | 52 | 99
    (all) | 256.1 (268.67) | 215.1 (231.74) | 234.5 (249.50)
Height [Mean (Standard Deviation); unit: cm] | 162.29 (10.151) | 160.87 (10.348) | 161.55 (10.227)
Weight [Mean (Standard Deviation); unit: kg] | 81.56 (21.948) | 82.50 (22.004) | 82.05 (21.871)
Number of Cardiovascular Risk Factors [Number; unit: participants]
  0 | 0 | 2 | 2
  1 | 7 | 1 | 8
  2 | 6 | 12 | 18
  >2 | 35 | 37 | 72
Homeostatic model assessment of insulin resistance (HOMA-IR) [Mean (Standard Deviation); unit: units on a scale] — HOMA-IR stands for "Homeostatic Model Assessment for Insulin Resistance" and it is calculated from fasting glucose and fasting insulin. HOMA-IR = (Insulin (mU/L) × Glucose (mg/dL)) / 405. Less than 1 means you are insulin-sensitive (optimal), greater than 1.9 indicates early insulin resistance, and greater than 2.9 indicates significant insulin resistance. Population: 6 participants did not have the HOMA-IR assessment completed at baseline and this was noted as a protocol deviation
  units on a scale
    number analyzed (Participants) | 45 | 49 | 94
    (all) | 3.42 (2.885) | 3.22 (2.297) | 3.32 (2.583)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.95 (7.837) | 32.03 (8.301) | 31.51 (8.059)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 96.90 (17.518) | 100.07 (19.128) | 98.56 (18.357)
Testicular adrenal rest tumor (TART) Volume [Mean (Standard Deviation); unit: mL] — Population: Only male participants with a history of TART had baseline value measured.
  mL
    number analyzed (Participants) | 8 | 5 | 13
    (all) | 2.1056 (2.32648) | 2.2170 (2.32177) | 2.1485 (2.22651)
Hospital Anxiety and Depression Scale (HADs) Total Score [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale (HADS) is a 14-item tool used to screen for anxiety (7 items) and depression (7 items). Each item is rated on a 4-point scale with 0 = none and 3 = very often. Scores for each of the 7 items (anxiety or depression) are calculated by adding together the values for each question; therefore, 21 is the highest score for either category (depression or anxiety). The total score for the combined anxiety and depression items (14 items total) is 42. Scores are interpreted as: 0-7 = normal; 8-10 = mild; 11-14 = moderate; and 15-21 = severe. Population: 1 participant did not have the HADs assessment completed at baseline and this was noted as a protocol deviation
  units on a scale
    number analyzed (Participants) | 48 | 51 | 99
    (all) | 8.1 (6.01) | 6.2 (4.90) | 7.2 (5.52)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Daily GC Dose in Subjects With Classic CAH Over the 24-week, Double Blind, Placebo-Controlled Treatment Period
Description: Absolute change from baseline (Day 1) in GC dose in HCe at Week 24. The analysis of absolute change in total daily GC dose in HCe will include data from Weeks 3, 6, 12, 18 and 24 in a mixed model
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Tildacerfont Group | Placebo
Number analyzed (Participants) | 48 | 52
mg | -5.0 (8.91) | -4.3 (9.75)

2. Secondary Outcome: Effect of Tildacrfont in Reducing GC Use to Near-physiologic Levels While Maintaining Androgen Control in Subjects With CAH
Description: Proportion of subjects with GC dose ≤11mg/m2/day in HCe and A4 ≤1.2x baseline or A4 ≤ ULN at Week 24
Time Frame: 24 weeks
Population: Responders are subjects with glucocorticoid dose ≤11 mg/m2/day in HCe and A4 ≤ 1.2x Baseline or A4 ≤ ULN at Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Tildacerfont Group | Placebo
Number analyzed (Participants) | 48 | 52
Participants | 4 | 5

3. Secondary Outcome: Effect of Tildacrfont in Reducing GC Use to Near-physiologic Levels While Maintaining Androgen Control in Subjects With CAH
Description: Proportion of subjects with baseline GC dose ≤ 35mg HCe who achieve GC dose ≤11 mg/m2/day in HCe and A4 ≤ 1.2x baseline or ≤ ULN at Week 24
Time Frame: 24 Weeks
Population: Responders are subjects with baseline glucocorticoid dose ≤ 35 mg HCe and glucocorticoid dose ≤11 mg/m2/day in HCe and A4 ≤ 1.2x Baseline or A4 ≤ ULN at Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Tildacerfont Group | Placebo
Number analyzed (Participants) | 19 | 25
Participants | 2 | 4

4. Secondary Outcome: Effectiveness in Reducing Cardiovascular Risk in Subjects With CAH
Description: Proportion of subjects with improvement in at least one cardiovascular risk factor at Week 24
Time Frame: 24 Weeks
Population: Responders are subjects with improvement in ≥ 1 baseline cardiovascular risk factor at Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Tildacerfont Group | Placebo
Number analyzed (Participants) | 48 | 50
Participants | 26 | 19

ADVERSE EVENTS:
Time Frame: The study period was expected to be up to 240 weeks in duration (double-blind treatment [24 weeks], open-label treatment [52 weeks], and optional open-label extension [up to the 240th week]), but due to early study termination, the total study period was 205 weeks. No subject entered the optional open label extension. The final safety follow-up was assessed at 30 days after the last dose of study drug for each participant.
Groups:
- Placebo: Placebo administered daily via oral tablet for 24 weeks
- Open Label Extension: Open label tildacerfont 200 mg for 52 weeks
Arm/Group | Tildacerfont Group | Placebo | Open Label Extension
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/52 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/52 | 2/92
Other Adverse Events (participants affected / at risk) | 11/48 | 16/52 | 77/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tildacerfont Group (N=48) | Placebo (N=52) | Open Label Extension (N=92)
adrenocortical insufficiency acute (Endocrine disorders) | 0 | 0 | 1
intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tildacerfont Group (N=48) | Placebo (N=52) | Open Label Extension (N=92)
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 5
Headache (Nervous system disorders) | 7 | 9 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3
Adrenal insufficiency (Endocrine disorders) | 3 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 5 | 7
Vomiting (Gastrointestinal disorders) | 3 | 6 | 11
Diarrhea (Gastrointestinal disorders) | 5 | 3 | 6
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 5
Fatigue (General disorders) | 6 | 8 | 16
Pyrexia (General disorders) | 3 | 2 | 3
Influenza like illness (General disorders) | 3 | 1 | 5
COVID-19 (Infections and infestations) | 6 | 5 | 9
Nasopharyngitis (Infections and infestations) | 5 | 2 | 17
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 7
Gastroenteritis (Infections and infestations) | 1 | 0 | 9
Influenza (Infections and infestations) | 2 | 1 | 5
Respiratory tract infection (Infections and infestations) | 0 | 1 | 5
Dizziness (Nervous system disorders) | 0 | 2 | 7
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 6

LIMITATIONS AND CAVEATS:
Due to early termination of the study, not all assessments were performed. Additionally, due to protocol deviations, some assessments and samples were not collected therefore data are not available for every assessment from every participant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT04544410/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/10/NCT04544410/SAP_001.pdf
  • Informed Consent Form (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT04544410/ICF_002.pdf